CLINICAL TRIAL: NCT05311449
Title: The Effect of Acupressure After Cesarean Section on Pain Intensity and First Mobilization Distance: A Double-Blind Randomized Controlled Study
Brief Title: The Effect of Post-Cesarean Section Acupressure on the Severity of Pain and First Mobilization Distance
Acronym: Acupress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mersin Universit
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pain; Mobilization
Keywords: Post-cesarean; Acupressure; Pain; Step; Mobilization
MeSH Terms: conditions — Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial, double blind
Masking Description: In the study, a researcher (T.Ç.Y.) will determine the acupressure and placebo points to be applied to women. However, the researcher (A.A.) who will apply acupressure and placebo acupressure be blinded without knowing whether these points are acupressure or placebo points. Participants will not know that they are in the acupressure or placebo group. Thus, the research will be carried out as a double-blind randomized controlled trial. When the research is completed, the data of the control and study groups (A or B) will be transferred to the computer environment by a researcher independent of the research, and the data will be analyzed by a statistician and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure Group (experimental) (Experimental): The experimental group will be given acupressure.
  Interventions: Other: Acupressure
- Placebo Acupressure Group (control) (Placebo Comparator): The placebo group will be given placebo acupressure.
  Interventions: Other: Plasebo acupressure

INTERVENTIONS:
Other: Acupressure — The experimental group will start with LI4 points, and continue with P6 and SP6 points. The application will be carried out by determining the priority order of the points with the draw. Attention will be paid to the intensity and duration of the pressure deemed appropriate. Since the individuals' responses will differ, the stiffness and pressure will be adjusted according to the individual's sensitivity not to cause tissue damage. Before starting the application, around the area to be pressed for 20-30 seconds will be gently rubbed with palm. With the gentle rubbing of the surrounding tissue, the tension and tissue sensitivity in warming, relaxing and preparatory will be reduced, and the tissue will be relieved. After, the point determined will be pressed manually for 2 minutes.
  Other Names: Acupress
  Arms: Acupressure Group (experimental)
Other: Plasebo acupressure — In the control group, the application will start with the points 1.5 cm around the LI4, P6 and SP6 points. The application process will continue in the same way with acupressure group and the pressure intensity will be less.
  Other Names: Placebo Acupress
  Arms: Placebo Acupressure Group (control)

SUMMARY:
This randomized controlled trial evaluates the effect of acupressure application on cesareans' pain and the number of steps in the first mobilization. This study hypothesizes that acupressure reduces pain and improves number of steps.

DETAILED DESCRIPTION:
Methods: In the study, 64 cesareans will randomly assigned to acupressure and placebo acupressure groups. To the acupressure group (n = 32), an average of 15 minutes will be applied to the LI4 (liver), P6 (pericardium) and the Sanyinjia points on the splenic meridian (SP6) located on the inner side of the lower leg, four fingers above the ankle and behind the tibia. In the placebo acupressure group (n = 32), the points 1.5 cm away from the LI4, P6 and SP6 points (four points in total) will be applied for an average of 15 minutes. The primary outcome of the research is the effect of acupressure on the pain of cesareans. The secondary outcome of the study is to determine the effect of acupressure on the number of steps. The pain will be collected before and 1 minute, 2nd and 4th hour after acupressure and placebo acupressure administration. The number of steps will be collected 4th hour after acupressure and placebo acupressure administration.

ELIGIBILITY:
Inclusion Criteria:

* Being conscious,
* The mother tongue is Turkish,
* To be oriented and cooperative,
* be between 18-45 years old,
* To voluntarily agree to participate in the study (signing the Informed Consent Form),
* Repeated cesarean section,
* Cesarean section under spinal anesthesia,
* Not having a risky pregnancy (preeclampsia, gestational diabetes etc.),
* No health problems of the fetus,
* To have given birth by cesarean section between 37-40 weeks,
* To be in the second hour of the postpartum period,
* Not receiving post-op patient-controlled analgesia,
* Not to have smoked or used alcohol during pregnancy,
* No complications in the mother and/or newborn after cesarean section,
* No sensitivity in the area where acupressure will be applied,
* Absence of any systemic or psychiatric diagnosis,
* Absence of active COVID-19 infection.

Exclusion Criteria:

* Lack of consciousness,
* The mother tongue is not Turkish,
* Not oriented and cooperative,
* Not to be between the ages of 18-45,
* Refusal to voluntarily participate in the study (those who did not sign the Informed Consent Form),
* Normal birth or cesarean delivery under general anesthesia,
* Cesarean delivery due to the risk of deterioration of maternal or fetal health,
* Not having had a risky pregnancy (preeclampsia, gestational diabetes, etc.),
* Not giving birth outside 37-40 weeks and by cesarean section,
* Not in the second hour of the postpartum period,
* Receiving post-op patient-controlled analgesia,
* To have used cigarettes and alcohol during pregnancy,
* Sensitivity in the area where acupressure will be applied,
* Presence of any systemic or psychiatric diagnosis,
* Active COVID-19 infection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the visual analog scale | Change from before implementation and after 1 minute, 2nd and 4th hour after implementation
  The total scale score is in the range of 0 cm (minimum) -10 cm (maximum). A score of 0 indicates no pain and a score of 10 indicates very severe pain.

SECONDARY OUTCOMES:
The number of steps using step counter (TNV 3D Pedometer (Model: PM2000, Made in China) | Change 4th hour after acupressure
  The number of steps in the first mobilization will be evaluated with a pedometer.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu VEFİKULUÇAY YILMAZ, Doctorate, Study Director — Mersin University; Aslıhan AKSU, master, Principal Investigator — Mersin University; Filiz DEĞİRMENCİ, master, Principal Investigator — Mersin University; Gülay ALTUN UĞRAŞ, doctorate, Principal Investigator — Mersin University; Mürşide ÇEVİKOĞLU KILLI, doctorate, Principal Investigator — Mersin City Hospital
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Xiang XY, Chin KHR, Gao J, Wu J, Lao L, Chen H. Acupressure for labor pain management: a systematic review and meta-analysis of randomized controlled trials. Acupunct Med. 2021 Aug;39(4):243-252. doi: 10.1177/0964528420946044. Epub 2020 Aug 18. PMID 32811182
- [Result] Smith CA, Collins CT, Levett KM, Armour M, Dahlen HG, Tan AL, Mesgarpour B. Acupuncture or acupressure for pain management during labour. Cochrane Database Syst Rev. 2020 Feb 7;2(2):CD009232. doi: 10.1002/14651858.CD009232.pub2. PMID 32032444
- [Result] Akgun M, Boz I. The effects of acupressure on post-cesarean pain and analgesic consumption: a randomized single-blinded placebo-controlled study. Int J Qual Health Care. 2020 Nov 16;32(9):609-617. doi: 10.1093/intqhc/mzaa107. PMID 32877509